CLINICAL TRIAL: NCT06733649
Title: Treatment Education for Pre- and Postpartum Women and Their Community Support
Brief Title: Treatment Education for Perinatal Women and Their Community Support
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB00478467
Record Dates: First submitted 2024-12-10; First posted 2024-12-13 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Opioid Dependency
Keywords: opioid dependence; perinatal women; social support
MeSH Terms: conditions — Opioid-Related Disorders

STUDY DESIGN:
Intervention Model Description: Perinatal women and the woman's community support will receive one treatment education session.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment education for perinatal women and the womens' community support (Experimental)
  Interventions: Other: substance abuse treatment education

INTERVENTIONS:
Other: substance abuse treatment education — Perinatal women and the women's community support will receive a 50 minute education session that provides correct information on opioid agonist medications and neonatal abstinence syndrome.

SUMMARY:
The study evaluates the feasibility and acceptability of a 50 minute treatment education session for perinatal women with opioid use disorder and a community support person. The education session provides correct information about opioid agonist medications and neonatal abstinence syndrome.

DETAILED DESCRIPTION:
Perinatal women with opioid disorder often face criticism by social network members for receiving opioid agonist treatment. Feeling stigmatized by others may impact willingness to start and remain in agonist treatment.

The present study evaluates the feasibility and acceptability of a 50 minute treatment education session for perinatal women who are treated using an agonist medication (methadone or buprenorphine) and community support chosen by the patient.

Study participants will be recruited from perinatal women who receive substance abuse treatment at the Center for Addiction and Pregnancy or Addiction Treatment Services at Johns Hopkins Bayview campus. These women will work with a counselor to select a community support person to bring to the program for the education session.

The session will provide correct information on opioid agonist medications and neonatal abstinence syndrome. This session will follow a structured outline.

ELIGIBILITY:
Inclusion Criteria:

* perinatal women treated with agonist medication
* interest in study participation
* interest in community support:
* interest in study participation

Exclusion Criteria:

* perinatal women not treated with agonist medication
* not interested in study participation
* not interested in community support:
* not interested in study participation

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2026-07-06 (Estimated); Primary Completion 2027-07-05 (Estimated); Study Completion 2027-12-05 (Estimated)

PRIMARY OUTCOMES:
Percentage of women interested in study participation | Immediately before session 1
  Feasibility -- percentage of women interested in study participation
Percentage of interested women who bring in community support to the education group | Immediately before session 1
  Acceptability -- proportion of interested women who bring in community support to the education group

SECONDARY OUTCOMES:
Knowledge as assessed by survey | Baseline, Immediately after session 1
  Women and the womens' community support will complete a 10 question true / false test before and after the education session

CONTACTS AND LOCATIONS:
Overall Officials: Michael Kidorf, Ph.D., Principal Investigator — Johns Hopkins University

IPD SHARING:
Plan to Share IPD: No